CLINICAL TRIAL: NCT02530801
Title: Management of Recurrent Pterygium to Prevent Visual Impairment
Brief Title: Strategies for Management of Recurrent Pterygium
Acronym: REPEAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15073
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Pterygium
MeSH Terms: conditions — Pterygium | interventions — Bevacizumab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin and 5 fluorouracil (Other): Subconjunctival injection of bevacizumab combined with 5 fluorouracil
  Interventions: Drug: Bevacizumab; Drug: 5 fluorouracil

INTERVENTIONS:
Drug: Bevacizumab — Subconjunctival injection of Bevacizumab combined with 5 fluorouracil in the recurrent pterygium
  Other Names: Avastin
Drug: 5 fluorouracil — Subconjunctival injection of Bevacizumab combined with 5 fluorouracil in the recurrent pterygium
  Other Names: ATC code: L01BC02

SUMMARY:
Pterygium is a common eye disease. Its mechanism remains unknown but studies suggest that it is related to exposure to ultraviolet rays and ocular dryness. Pterygium affects vision by causing astigmatism and may encroach on cornea (transparent part of the eye) affecting vision. It could cause ocular irritation and can be cosmetically unacceptable especially when inflamed.

Recurrence is the most common outcome of pterygium excision. Recurrence rates of pterygium vary from 10 to more than 80%. Recurrence can be detected first in the conjunctiva(skin of your eye), before advancing on to the cornea. Treating the recurrent pterygium before the cornea gets involved avoids repeat surgery, which is difficult and is associated with more scarring. To avoid repeated surgeries, the activity of a recurrent pterygium should be stopped before it progresses to true recurrence.

Several studies attributed the recurrence pf pterygium to the increase of substances as vascular endothelial growth factor(VEGF) and fibroblast growth factor. Avastin (Anti-VEGF) and 5 fluorouracil(5FU) (antimetabolite) are medications that suppress the formation of VEGF and fibroblast growth factor.

Studies have shown that the subconjunctival injection of 5 F and Avastin into the recurring pterygium has been both safe and effective in treatment of recurrent pterygium.

In many cases, vascularization and inflammation were controlled by subconjunctival Avastin, providing evidence for a role of VEGF in pterygium formation. 5FU is widely used in ophthalmology because of its anti-scarring properties.

The other option for treatment of recurrent pterygium is surgery. Recurrent pterygium is a challenging condition that usually resists conventional surgery and its rate of recurrence after surgery is high. Moreover, recurrent pterygium surgery is usually accompanied by scarring, more risk of intra and post- complications This study aims to generate data to inform further studies towards establishing Avastin and 5 fluouracil as treatment modality for recurrent pterygium.

DETAILED DESCRIPTION:
Purpose To assess the efficacy of combined 5FU and Avastin injections in the treatment of recurrent pterygium.

Design Pilot study. The patients will receive combined 5FU and Avastin injection.

Methodology Patients for inclusion in the study will be identified in the specialist corneal clinics at Queens Medical Centre.

5 FU injection

Dose: 0.15 ml of 5FU (3.75mg) will be administered into the body of the recurring pterygium up to 5 injections as determined by response. The 5FU solution is prepared locally in the pharmacy for ophthalmic use. It will be delivered preloaded in a 1ml syringe containing 0.3 ml of 2.5mg 5FU per 0.1ml. The injection will be given under topical anaesthesia. One to two drops of 5% povidone iodine will be instilled in the conjunctival sac 5min before the injection. All injections will be given in the outpatient clinic using a slit lamp. The needle (27Gauge) will be advanced in a zigzag manner into the subconjunctival space, avoiding any large blood vessels, until the middle of the lesion is reached. The solution will be then injected and the needle withdrawn. After the injection, 1-2 drops of chloramphenicol 0.5% preservative free minims will be instilled topically and continued four times a day for 3 days after each injection. Injections will be carried out every two weeks as described above. Patients will have the ability to access the 24 hour on call emergency eye service, and at the same time be provided with contact numbers for investigators for any queries during the study period.

Avastin injection

Dose: 0.15 ml of Avastin (2.5 mg/0.1 ml) will be administered in the body of the recurrent lesion. Up to 5 injections could be given.

The injection will be given under topical anaesthesia. One to two drops of 5% povidone iodine will be instilled in the conjunctival sac 5min before the injection. All injections will be given in the outpatient clinic using a slit lamp. The needle (27Gauge) will be advanced in a zigzag manner into the subconjunctival space, avoiding any large blood vessels, until the middle of the lesion is reached. The solution will be then injected and the needle withdrawn. After the injection, 1-2 drops of chloramphenicol 0.5% preservativefree minims will be instilled topically and continued four times a day for 3 days after each injection. Injections will be carried out every two weeks as described above. Patients will have the ability to access the 24 hour on call emergency eye service, and at the same time be provided with contact numbers for investigators for any queries during the study period.

Fluorescein angiography (FFA) will be done to characterise the conjunctival vessels. It is a safe routine investigation that is done on daily basis in eye clinics.

Patient Inclusion Criteria will be:

* Patients over the age of 18
* Able to give informed consent
* Patients with recurrent pterygium within 6 months of original excision[Recurrence is defined in the protocol (page 22)]
* Use of effective contraception in females of childbearing age

Patient exclusion criteria will be:

* Patients under 18 years of age
* Patients unable or refusing to provide informed consent
* Patients who are needle phobic
* Pregnant women, women aiming for conception and breast feeding women.
* Patients with hypersensitivity to the active substance or to any of the excipients
* Patients with active or suspected ocular or periocular infections.
* Patients with active severe intraocular inflammation.
* Patients with raised intraocular pressure or on glaucoma medication
* Patients with advanced recurrent pterygium that extends between the pupil and limbus at the time of presentation

In case of bilateral eye involvement, only one eye will be treated with the study drug. The study participants will reserve the right to withdraw from the study at any stage, and will be kept up to date with any new information available about the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients able to give informed consent- Patients with early recurrent pterygium within 6 months of original excision (conjunctival recurrence or recurrence extending just across the limbus).
* Use of effective contraception in females of childbearing age.

Exclusion Criteria:

* Patients under 18 years of age
* Patients unable or refusing to provide informed consent
* Patients who are needle phobic
* Pregnant women, women aiming for conception and breastfeeding women
* Patients with hypersensitivity to the active substance or to any of the excipients
* Patients with active or suspected ocular or periocular infections.
* Patients with active severe intraocular inflammation.
* Patients with raised intraocular pressure or on glaucoma medication
* Patients with advanced recurrent pterygium that extends between the pupil and limbus at the time of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Arrest of progression of the fibrovascular tissue will be measured using slit lamp (width of the lesion in millimeters) | At 3 month, which is 2 weeks after the last injection
  The width of the lesion will be measured on slit lamp in millimeters

SECONDARY OUTCOMES:
Disappearance of redness of the lesion will be assessed using the slit lamp | At 3 month, which is 2 weeks after the last injection
  Images will be taken using anterior segment slit lamp camera and will be compared for redness by 2 different observers
Return of conjunctiva to normal thickness will be measured using slit lamp (millimeters) | At 3 month, which is 2 weeks after the last injection
  The thicknessof the lesion will be measured on slit lamp in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Harminder Dua, Professor, Principal Investigator — University of Nottingham

REFERENCES:
- [Background] Said DG, Faraj LA, Elalfy MS, Yeung A, Miri A, Fares U, Otri AM, Rahman I, Maharajan S, Dua HS. Intra-lesional 5 fluorouracil for the management of recurrent pterygium. Eye (Lond). 2013 Oct;27(10):1123-9. doi: 10.1038/eye.2013.135. Epub 2013 Jun 28. PMID 23807385